CLINICAL TRIAL: NCT03489694
Title: Within-tester Repeatability and Between-tester Reproducibility of Skin Test Endpoint Titration
Brief Title: Repeatability and Reproducibility of Skin Test Endpoint Titration
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, College of Medicine, University of Saskatchewan
Other Study IDs: STE-2018
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Allergic Reaction
Keywords: skin test endpoint
MeSH Terms: conditions — Hypersensitivity | interventions — Skin Test End-Point Titration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Each subject will undergo skin test endpoint titrations with three different testers.
  Interventions: Procedure: Skin test endpoint titration

INTERVENTIONS:
Procedure: Skin test endpoint titration — An allergen that is suitable to cause skin reactions when introduced to the forearm through pricking will be administered in doubling concentrations.

SUMMARY:
This study will examine the within-tester repeatability and between-tester reproducibility of skin test endpoint titrations performed in those with allergic sensitivities.

DETAILED DESCRIPTION:
Participants will be recruited from the local community. Participants with a previous history of skin prick testing in our lab will not be required to undergo preliminary skin prick testing, as the allergen to be used for skin prick titrations is known. New participants will undergo skin prick testing. The procedures for skin prick testing and skin test endpoint (STE) titration will be guided by the AllerGen CIC Allergen Skin Titration by Epicutaneous Method (Prick) Standard Operating Procedure. Different allergen extracts for the skin prick test or different doubling doses of an allergen in duplicate for the STE will be applied to the forearm, pricked with a lancet, and assessed ten minutes later by measuring the wheal sizes produced. The study will require three visits to the lab (i.e. three testers), each separated by one week and lasting roughly 30 minutes. Each visit will entail the duplicate STE procedure performed by a different tester. If a participant is new to the lab, they will undergo skin prick testing during their first lab visit prior to undergoing the skin prick titration and so, their first study visit may last up to one hour.

ELIGIBILITY:
Inclusion Criteria:

* must have allergic sensitivities confirmed by a skin prick test (or historically) to at least one of the study allergens

Exclusion Criteria:

* skin condition on the forearms
* if there is a situation where interpretation of skin reactions would be difficult (e.g. sleeve tattoos, scarring)
* regular use of anti-histamines (assessed on a case-by-case basis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Within-tester repeatability | 10 minutes post skin pricking
  Comparison of wheal size (in mm) of skin reactions caused by a tester (duplicate skin pricking for each concentration of allergen administered)
Between-tester reproducibility | approximately 3 weeks (one week washout between tests)
  Comparison of wheal size (in mm) of skin reactions caused by three different testers

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blais CM, Davis BE, Cockcroft DW. Within-tester repeatability and between-tester reproducibility of skin test endpoint titration: A quality assurance study. Ann Allergy Asthma Immunol. 2019 Feb;122(2):220-222. doi: 10.1016/j.anai.2018.10.009. Epub 2018 Oct 14. No abstract available. PMID 30326324